CLINICAL TRIAL: NCT04372823
Title: Promoting Nutrition and Physical Activity in Family Child Care
Acronym: FCCH
Status: Completed | Type: Observational
Sponsor: University of South Carolina (Other)
Collaborators: Johns Hopkins University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Russell Pate, Professor, University of South Carolina
Other Study IDs: Pro00066175; R01HD093784 (NIH)
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Diet, Healthy; Physical Activity; Obesity, Childhood
MeSH Terms: conditions — Motor Activity; Pediatric Obesity | interventions — Policy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Comparison: Comparison children within family child care homes not exposed to policy/program
- Intervention: Intervention children within family child care homes exposed to policy/program
  Interventions: Behavioral: Policy/program

INTERVENTIONS:
Behavioral: Policy/program — Policy/program to improve nutrition and increase physical activity
  Groups: Intervention

SUMMARY:
The CHEER study takes advantage of a natural experiment happening in South Carolina (SC). The South Carolina Department of Social Services implemented new healthy eating and physical activity standards through a state-wide policy for family child care homes that participate in the ABC Grow Healthy program. Thus, CHEER is a quasi-experimental, two-group, pre-test/post-test design study.

DETAILED DESCRIPTION:
The overall goal of the study is to evaluate new healthy eating and physical activity standards targeting family child care homes in South Carolina. To accomplish this goal, we are assessing the effects of the standards on the dietary intake and physical activity levels of racially diverse low-income children in family child care homes. The specific aims of the "CHEER" study are as follows:

Aim 1. Evaluate the extent to which the new regulatory standards impact children's dietary intake assessed via direct observation in homes and 24-hour recalls with parents, and physical activity and sedentary behavior assessed via accelerometry.

Aim 2. Evaluate the extent to which the new regulatory standards impact children's body mass index computed from researcher-measured height and weight.

Secondary Aim. Evaluate the extent to which family child care homes in the SC ABC Child Care Program comply with the new healthy eating and physical activity regulatory standards, compared to family child care homes not participating in the program.

We hypothesize that most homes will comply with the new standards, yielding improvements in children's healthy eating and physical activity levels. As an exploratory aim, we will examine the effects of the standards on children's weight status.

ELIGIBILITY:
Inclusion Criteria:

* Having a child in care between the ages 2 and 4 years at recruitment
* The family is planning to stay in the same care arrangement for the next few years

Exclusion Criteria:

* Family planning to leave the care arrangement in next few years

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Family child care homes located in South Carolina and children ages 2-4 years enrolled in those homes.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Diet | Approx 1 year
  Healthy Eating Index score - The Healthy Eating Index is a calorie-adjusted comparison of individual or group-level dietary intake to current dietary guidelines. The Healthy Eating Index was last updated in 2015 and represents the sum of thirteen component scores. Higher scores are awarded for healthier intake within each component. Each component of the Healthy Eating Index has a standard for receiving the minimum or maximum points possible. The HEI components and maximum scores include: total fruit (5), whole fruit (5), total vegetables (5), greens and beans (5), whole grains (10), dairy (10), total proteins (5), seafood/plant (lean) proteins (5), fatty acids (10), refined grains (10), sodium (10), added sugars (10), and saturated fats (10).
Physical activity | Approx every year for 2 years
  Accelerometer measured minutes of moderate to vigorous physical activity

SECONDARY OUTCOMES:
Body mass index | Approx every year for 2 years
  Child body mass index z-score
Family child care home environment | Approx every year for 2 years
  Environment and Policy Assessment and Observation

CONTACTS AND LOCATIONS:
Overall Officials: Russell R Pate, Principal Investigator — University of South Carolina
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - University of South Carolina, Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: No